CLINICAL TRIAL: NCT06606184
Title: Benefits of Pulmonary Rehabilitation to Patients Post Liver Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Collaborators: Chang Gung University of Science and Technology (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hui-Ling Lin, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202102058B0
Record Dates: First submitted 2024-09-16; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Liver Transplant Surgery
Keywords: liver transplant; pulmonary rehabilitation; inspiratory muscle training; inspiratory muscle strength; Dyspnea
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inspiratory Muscle Training group (Experimental): Participants received a 12-week inspiratory muscle training and incentive spirometry therapy after discharged from hospital
  Interventions: Procedure: Inspiratory muscle Training
- Routine care (Sham Comparator): Participants received incentive spirometry therapy only
  Interventions: Procedure: Routine Care

INTERVENTIONS:
Procedure: Inspiratory muscle Training — Participants underwent a 12-week program consisting of inspiratory muscle training twice daily, incentive spirometry three times daily, and upper limb exercises along with marching in place for 30 minutes.
  Arms: Inspiratory Muscle Training group
Procedure: Routine Care — Participants received routine care, which included encouragement to use incentive spirometry three times daily.
  Arms: Routine care

SUMMARY:
The goal of this clinical trial was to access the benefits of a 12-week home-based pulmonary rehabilitation regimen on pulmonary function recovery in post-liver transplant patients. The main questions it aims to answer are:

Does pulmonary rehabilitation facilitate pulmonary muscle strength recovery? Does the intervention improve pulmonary function and reduce dyspnea sensation?

Participants performed:

Inspiratory muscle training twice a day for 12 weeks after discharged from the hospital Upper limb resistive training Lower limb exercise

DETAILED DESCRIPTION:
Patients undergoing liver transplantation often face significant challenges related to pulmonary rehabilitation. Although postoperative rehabilitation has been extensively studied, the specific role of pulmonary rehabilitation programs has received limited attention. This study aims to evaluate the efficacy of a home-based pulmonary rehabilitation program in improving respiratory function recovery among post-liver transplant patients. The training group participated in a 12-week pulmonary rehabilitation program post-discharge, emphasizing respiratory muscle and exercise training, while the control group received standard care, which included traditional rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 years or older
* Scheduled to undergo living donor liver transplantation
* Stable vital signs
* Normal cognitive function
* Able to perform activities independently using their own strength and coordination
* Willing and able to participate in 12 weeks of rehabilitation training

Exclusion Criteria:

* Severe physical illness during the operation
* Acute bleeding
* Unstable vital signs
* Hepatic encephalopathy, or neurological conditions such as stroke, Parkinson's disease, or cognitive dysfunction
* Limited mobility (e.g., unable to stand, lift upper limbs, or bedridden)
* Inability to comply with 12 weeks of pulmonary rehabilitation post-discharge
* Unstable vital signs
* Hepatoencephalopathy, such as cardiovascular accident, Parkinson disease, cognitive dysfunction
* Those with limited mobility (unable to stand, unable to lift upper limbs, or bedridden)
* Those who are unable to cooperate with the 12 weeks of pulmonary rehabilitation exercises after discharge.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Respiratory Muscle Stregnth Test | Throughout the study completion, approximately 3 month
  Respiratory muscle strength was determined by Maximum Inspiratory Pressure (MIP) using a pressure monometer.

SECONDARY OUTCOMES:
Oxygenation status | Participants underwent maximum inspiratory and expiratory pressure measurements at four time points: upon admission, before discharge from the intensive care unit, before discharge from the hospital, and at the end of the 12-week enrollment period.
  Oxygen saturation was monitored using a pulse oximeter.
Dyspnea Severity Assessment | Throughout the study completion, approximately 3 month
  Dyspnea severity was assessed by a rating of perceived exertion, using the Borg Scale which ranged from 0 (no respiratory difficulty) to 10 (extreme respiratory difficulty), with higher scores indicating more severe breathing difficulty.
Forced Vital Capacity | Throughout the study completion, approximately 3 month
  The forced vital capacity was obtained, using spirometry, by having the patient take a deep breath and then exhale forcefully. The test results were based on three reproducible measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Jui-Fang Lin, PhD, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The data is available upon request from the principal investigator.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 3 three years after the study is completed.
Access Criteria: The data is available upon request from the principal investigator.

REFERENCES:
- [Background] Au KP, Chan SC, Chok KS, Sharr WW, Dai WC, Sin SL, Wong TC, Lo CM. Clinical factors affecting rejection rates in liver transplantation. Hepatobiliary Pancreat Dis Int. 2015 Aug;14(4):367-73. doi: 10.1016/s1499-3872(15)60391-5. PMID 26256080
- [Background] Aamir,T., Iftikhar,S., Khan, R.R., &Khan, M.K (2019).Role of physiotherapy in improving quality Of life in liver transpant patients. The Rehabilitation Journal, 3(2),126-130.